CLINICAL TRIAL: NCT04256226
Title: Far Eastern Memorial Hospital
Brief Title: Clinical Outcome of Female Non-gastric Gastrointestinal Stromal Tumor
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 108174-E
Record Dates: First submitted 2020-02-04; First posted 2020-02-05 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-03

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tumor excision — Excision of GIST

SUMMARY:
To elucidate the prognosis of women with non-gastric primary gastrointestinal stromal tumors.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumor (GIST) are mesenchymal tumors arising from gastrointestinal tract, mesentery, or omentum. They took up about 3% of gastrointestinal malignancies. Although rarely, the clinical presentation of non-gastric GIST might mimick ovarian cancer, and would be managed by gynecologists. Therefore, retrospective review of female non-gastric GIST cases will be performed to investigate the clinical outcome of non-gastric GIST. The result of this study might be used as an important reference for gynecologists.

ELIGIBILITY:
Inclusion Criteria:

* > 20 years of women.
* non-gastric gastrointestinal stromal tumor

Exclusion Criteria:

* Those without pathological report or surgical record.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: non-gastric gastrointestinal tumor in women
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 20 years
  The date of surgery to the date of death or last follow-up

SECONDARY OUTCOMES:
Recurrence-free survival | 20 years
  The date of surgery to the date of recurrence or last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan